CLINICAL TRIAL: NCT06985069
Title: Impact of Multimodal Versus Opioid-Only Anesthesia on Short Term Quality of Recovery After Major Surgery: A Randomized Prospective Single-Center Superiority Trial
Brief Title: Outcome of Multimodal Anesthesia Bern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMA 25-01; 2025-00283 (Other: Business Administration System for Ethics Committees (BASEC))
Record Dates: First submitted 2025-05-06; First posted 2025-05-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use; Pain, Postoperative; Postoperative Complications; Postoperative Nausea
Keywords: Multimodal anesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, double-blind (patients and outcome assessment), superiority, two-arm controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal anesthesia-group (Experimental): The intervention consists of the application of a standardized combination of Magnesium, Ketamine, Lidocaine and Dexmedetomidine before and during surgery in combination with opioids (Fentanyl, Methadone, and Hydromorphon) in a non-standardized fashion for perioperative pain control.
  Interventions: Procedure: General anesthesia applying multimodal anesthesia
- Opioid based-group (Active Comparator): Patients in the control group will be treated with opioids only (Fentanyl, Methadone, Hydromorphone) at the discretion of the treating anesthetist for perioperative pain control.
  Interventions: Procedure: General anesthesia using conventional opioid-based regimen

INTERVENTIONS:
Procedure: General anesthesia applying multimodal anesthesia — In the multimodal anesthesia-group a combination of different opioid-sparing drugs are added for general anesthesia, dosages are as follows:
  * Magnesium 2g IV
  * Dexmedetomidine IV 0.3mcg/kg IBW bolus over 10 minutes, followed by 0.3mcg/kg IBW until 30 min. before the end of surgery or the maximal dosage of 1.4mcg/kg IBW.
  * Ketamine IV 0.3mg/kg IBW bolus, followed by 0.3 mg/kg IBW or a max. Dose of 25mg/h, until 30 min. before the end of surgery.
  * Lidocaine IV 1mg/kg IBW bolus, followed by 1mg/kg/h IBW until in PACU/ICU
  Arms: Multimodal anesthesia-group
Procedure: General anesthesia using conventional opioid-based regimen — Opioids (Fentanyl, Methadone, Hydromorphone) at the discretion of the treating anesthetist
  Arms: Opioid based-group

SUMMARY:
In the context of the ongoing opioid crisis in the USA and Europe, reducing perioperative opioid use is a growing priority. Multimodal anesthesia (MMA) offers a patient-centered alternative to opioid-free anesthesia, combining regional techniques, non-opioid analgesics, and adjunct therapies to enhance pain control while minimizing opioid reliance. By targeting multiple pain pathways, MMA can improve recovery outcomes, reduce side effects, and optimize resource use, representing a potential paradigm shift in perioperative medicine.

This study compares (patient-centered) outcomes after application of MMA (a standardized combination of Magnesium, Ketamine, Lidocain and Dexmedetomidine before and during surgery in combination with opioids) with an opioid based general anesthesia regimen in the context of major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Existing informed consent
* German, Italian or French speaking
* Age 18 or more
* Planned duration of surgery 60min or more
* Inpatients and postoperative transfer to PACU or 24h ICU

Exclusion Criteria:

* Palliative or emergency procedures
* Reoperation (e.g. 2nd look)
* Bariatric surgery patients
* Pregnancy / breastfeeding
* Adults legally protected
* Known allergy or contraindication to interventional medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Patient centered satisfaction measured by the QoR-15 (Quality of Recovery-15 questionnaire with 15 questions) | Postoperative day 1
  QoR-15 is a score from 0 to 150 with higher scores corresponding to greater patient satisfaction

SECONDARY OUTCOMES:
Evolution of Patient centered satisfaction measured by the QoR-15 (Quality of Recovery-15-questionnaire) | Postoperative day 2
  QoR-15 is a score from 0 to 150 with higher scores corresponding to greater patient satisfaction
Safety outcome 1a respiratory: respiratory rate | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with reported respiratory rate of less than 8 per minute
Safety outcome 1b respiratory: airway obstruction needing an intervention | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with reported airway obstruction needing an intervention (e.g. insertion of a naso-pharyngeal-tube)
Safety outcome 1c respiratory: desaturation | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with reported desaturation (peripheral oxygen saturation < 92%) despite administration of nasal oxgen (max. 6l/min.)
Safety outcome 2a cardiac: hypotension | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with reported hypotension needing an intervention
Safety outcome 2b cardiac: bradycardia | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with reported heart rate lower than 60 beats per minute needing an intervention
Safety outcome 2c cardiac: conduction block | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Number of patients with a postoperatively new reported conduction block
Postoperative data 1: pain scores measured by numeric rating scale (NRS) | At arrival and after 6 hours/before leaving post-anesthesia care unit (PACU, expected up to 1 day) or intermediate care (IMC)
  NRS ranging from 0 to 10, with higher scores corresponding to more postoperative pain
Postoperative data 2: sedation score & delirium rate measured by the Richmond Agitation-Sedation Scale (RASS) | Maximal values during stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  RASS ranging from -5 until +4 with negative values corresponding to progressive sedation, positive values corresponding to progressive delirium
Postoperative data 3: severity of postoperative nausea and vomiting | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  percentage of patients with either:
  * no nausea
  * nausea without vomiting
  * nausea with vomiting
  * >3 times vomiting in 30 minutes
Postoperative data 4: oxygen use | During stay in post-anesthesia care unit (PACU) or intermediate care IMC (expected to be) up to 1 day
  Maximal administered oxygen ([l/min.]
Opioid consumption in the post-operative period | First 48 hours postoperatively
  Oral morphine milligram equivalents mg
Impact on long-term opioid use after hospital discharge | Hospital discharge (expected up to 3 weeks)
  Percentage of patients with a new opioid prescription after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wüthrich, Professor, Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital, Bern, Switzerland
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No